CLINICAL TRIAL: NCT04783285
Title: Effect of Individual Cognitive Stimulation at Home in Adults With Psychotic Disorders: Randomised Controlled Trial
Brief Title: Effect of Individual Cognitive Stimulation at Home in Adults With Psychotic Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CEDIARA - Assoc. Solidariedade Social de Ribeira de Fráguas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20210218
Record Dates: First submitted 2021-03-01; First posted 2021-03-05 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2021-02

CONDITIONS: Psychotic Disorders; Schizophrenia; Schizoaffective Disorder; Delusional Disorder; Substance-Induced Psychotic Disorder
Keywords: cognition; mood; executive functions; quality of life; non-pharmacological therapy; randomised controlled trial; schizophrenia; psychotic disorders; cognitive stimulation
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Schizophrenia, Paranoid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants who meet the inclusion criteria will be randomly assigned to the intervention group receiving CS or to a control group receiving treatment as usual. Participants in the intervention group will participate in two CS sessions per week for 16 weeks besides their treatment as usual. The sessions will be based on the existing protocol.
  Interventions: Behavioral: Individual cognitive stimulation therapy (iCST)
- Control Group (No Intervention): Participants assigned to the control group will maintain their usual treatment: social interaction activities, stimulation of personal skills, and any prescribed psychotic-specific medication.

INTERVENTIONS:
Behavioral: Individual cognitive stimulation therapy (iCST) — The intervention group will receive 32 individual CS sessions per participant. Each session will last approximately 45 minutes and will have the following structure: session introduction (5 minutes); reality orientation (10 minutes); stimulation of cognitive domain (25 minutes); session closure (5 minutes). The sessions will be led by a previously trained therapist. The intervention program will include several activities based on the principles of CS and adjusted for participants with psychotic disorders.
  Arms: Intervention Group

SUMMARY:
The aim of this study is to test the effect of cognitive stimulation (CS), applied individually and at home, on the overall cognitive functioning, emotional state, functionality, and quality of life (QoL) in adults with psychotic disorders. To this end, a randomised controlled clinical trial will be conducted in which selected participants will be randomly assigned to an individual intervention group using CS or a control group. The CS program is adapted from other existing protocol, composed of 32 sessions. Each session will last 45 minutes and will be held twice weekly. There will be four evaluation points (baseline, intra-evaluation - after 8 weeks of intervention, post-evaluation - after 16 weeks of intervention, follow-up - after 8 weeks of the end of intervention).

DETAILED DESCRIPTION:
Epidemiological studies indicate that Portugal has one of the highest prevalence rates of mental disorders in Europe. In 2016, one in five Portuguese suffered from a psychiatric illness and the network of Integrated Continuous Care in mental health is small, which is a major constraint to rehabilitation and support responses for people with mental health problems.

It is important to include psychologists and neuropsychologists in multidisciplinary teams, in actions related to mental health promotion and mental illness prevention programs, so that they can provide more comprehensive interventions for other effects of chronic mental health conditions, such as cognitive decline.

There is evidence linking psychotic disorders to impairments in functioning in most cognitive domains, including memory, executive functions, and attention, and that cognitive ageing in some areas may be accelerated in individuals with psychotic disorders. Thus, it is important to focus interventions on cognitive functioning in patients with psychosis, even after acute psychotic symptoms have improved. Executive functions appear to be of particular importance in the context of mental health problems, as they appear to be particularly integral for psychosocial functioning and the completion of instrumental activities of daily living. There is evidence that CS interventions in individual format are associated with greater effectiveness.

Many studies have supported the effectiveness and accessibility of home-based interventions in people with chronic mental illness. Yet, there are few published studies on continuous intervention in people with chronic mental illness and even more limited knowledge of how cognitive stimulation can help chronic mental health patients, including those with psychosis, to function.

One Portuguese study about the effect of an individual CS program in a home setting on cognitive and mood functioning in adults with psychotic disorders was tested, showed encouraging results and presented in detail an intervention protocol. However, it also presents some important limitations (e.g., convenience sample, lack of follow-up evaluation).

This study aims to overcome those limitations, through a randomised controlled trial, and, in addition to testing the effect of the CS program on global cognition, it also aims to assess its effect on emotional state, daily functioning, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adults under 65 years.
* Diagnosed with of schizophrenia spectrum and other psychotic disorders according to the criteria of DSM-5 (APA, 2013), determined by a professional clinician.
* Willing to participate in all intervention and assessment sessions.
* Provided informed consent.
* Native speakers of Portuguese.

Exclusion Criteria:

* Presentation of a condition requiring immediate intervention (e.g., suicidal thoughts).
* Severe sensory and physical limitations that prevent participation in the sessions.
* Severe disconnection with the environment and very limited attentional level.
* Inability to communicate adequately.
* Psychoactive substance use.
* Currently participating in another study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Cognitive functioning evaluated through Montreal Cognitive Assessment [MoCA] | baseline
  Cognitive functioning is assessed using the MoCA which is a brief cognitive screening. Scores range from 0 to 30, with higher scores indicating better cognitive functioning.
Change in cognitive functioning evaluated through MoCA | 8 weeks after the beginning of the intervention
  Cognitive functioning is assessed using the MoCA which is a brief cognitive screening. Scores range from 0 to 30, with higher scores indicating better cognitive functioning.
Change in cognitive functioning evaluated through MoCA | 16 weeks after the beginning of the intervention
  Cognitive functioning is assessed using the MoCA which is a brief cognitive screening. Scores range from 0 to 30, with higher scores indicating better cognitive functioning.
Change in cognitive functioning evaluated through MoCA | 8 weeks after end of intervention
  Cognitive functioning is assessed using the MoCA which is a brief cognitive screening. Scores range from 0 to 30, with higher scores indicating better cognitive functioning.
Executive functions evaluated through Frontal Assessment Battery (FAB) | baseline
  The FAB is used to assess executive function in several subtests: conceptualization, mental flexibility, motor programming, sensitivity to interference, inhibitory control, and environmental autonomy. Scores range from 0 to 18, with higher scores indicating better executive functioning.
Change in executive functions evaluated through FAB | 8 weeks after the beginning of the intervention
  The FAB is used to assess executive function in several subtests: conceptualization, mental flexibility, motor programming, sensitivity to interference, inhibitory control, and environmental autonomy. Scores range from 0 to 18, with higher scores indicating better executive functioning.
Change in executive functions evaluated through FAB | 16 weeks after the beginning of the intervention
  The FAB is used to assess executive function in several subtests: conceptualization, mental flexibility, motor programming, sensitivity to interference, inhibitory control, and environmental autonomy. Scores range from 0 to 18, with higher scores indicating better executive functioning.
Change in executive functions evaluated through FAB | 8 weeks after end of intervention
  The FAB is used to assess executive function in several subtests: conceptualization, mental flexibility, motor programming, sensitivity to interference, inhibitory control, and environmental autonomy. Scores range from 0 to 18, with higher scores indicating better executive functioning.

SECONDARY OUTCOMES:
Self-maintaining and instrumental activities of daily living evaluated through Lawton Instrumental Activities of Daily Living (IADL) Scale | baseline
  Lawton IADL Scale assesses level of independence of the elderly in relation to instrumental activities of daily living. A score is assigned according to the subject's ability to perform a given task. The score ranges between 8 and 30 points. The highest score corresponds to a higher degree of dependence.
Change in self-maintaining and instrumental activities of daily living evaluated through Lawton IADL Scale | 8 weeks after the beginning of the intervention
  Lawton IADL Scale assesses level of independence of the elderly in relation to instrumental activities of daily living. A score is assigned according to the subject's ability to perform a given task. The score ranges between 8 and 30 points. The highest score corresponds to a higher degree of dependence.
Change in self-maintaining and instrumental activities of daily living evaluated through Lawton IADL Scale | 16 weeks after the beginning of the intervention
  Lawton IADL Scale assesses level of independence of the elderly in relation to instrumental activities of daily living. A score is assigned according to the subject's ability to perform a given task. The score ranges between 8 and 30 points. The highest score corresponds to a higher degree of dependence.
Change in self-maintaining and instrumental activities of daily living evaluated through Lawton IADL Scale | 8 weeks after end of intervention
  Lawton IADL Scale assesses level of independence of the elderly in relation to instrumental activities of daily living. A score is assigned according to the subject's ability to perform a given task. The score ranges between 8 and 30 points. The highest score corresponds to a higher degree of dependence.
Depressive symptomatology assessed through the Center for Epidemiologic Studies Depression Scale (CES-D) | baseline
  This instrument evaluated depressive symptoms using 20 answers. Scores range between 0 and 60 points. Higher scores indicate more severe depressive symptoms.
Change in depressive symptomatology assessed through the CES-D | 8 weeks after the beginning of the intervention
  This instrument evaluated depressive symptoms using 20 answers. Scores range between 0 and 60 points. Higher scores indicate more severe depressive symptoms.
Change in depressive symptomatology assessed through the CES-D | 16 weeks after the beginning of the intervention
  This instrument evaluated depressive symptoms using 20 answers. Scores range between 0 and 60 points. Higher scores indicate more severe depressive symptoms.
Change in depressive symptomatology assessed through the CES-D | 8 weeks after end of intervention
  This instrument evaluated depressive symptoms using 20 answers. Scores range between 0 and 60 points. Higher scores indicate more severe depressive symptoms.
Quality of life (QoL) evaluated through World Health Organization Quality of Life-Bref (WHOQOL-BREF) | baseline
  The WHOQOL-BREF is used to assess QoL. Consisting of 26 items, it assesses several domains: physical health, mental health, social relationships and environment. The first 2 items are intended to assess the individual's perception of his/her general QoL and general health. The global score range between 0 to 100. Higher scores indicate better QoL perceived by the subject.
Change in QoL evaluated through WHOQOL-BREF | 8 weeks after the beginning of the intervention
  The WHOQOL-BREF is used to assess QoL. Consisting of 26 items, it assesses several domains: physical health, mental health, social relationships and environment. The first 2 items are intended to assess the individual's perception of his/her general QoL and general health. The global score range between 0 to 100. Higher scores indicate better QoL perceived by the subject.
Change in QoL evaluated through WHOQOL-BREF | 16 weeks after the beginning of the intervention
  The WHOQOL-BREF is used to assess QoL. Consisting of 26 items, it assesses several domains: physical health, mental health, social relationships and environment. The first 2 items are intended to assess the individual's perception of his/her general QoL and general health. The global score range between 0 to 100. Higher scores indicate better QoL perceived by the subject.
Change in QoL evaluated through WHOQOL-BREF | 8 weeks after end of intervention
  The WHOQOL-BREF is used to assess QoL. Consisting of 26 items, it assesses several domains: physical health, mental health, social relationships and environment. The first 2 items are intended to assess the individual's perception of his/her general QoL and general health. The global score range between 0 to 100. Higher scores indicate better QoL perceived by the subject.
Quality of life (QoL) evaluated through MOS Short Form Health Survey 36 Item v2 (SF-36v2) | baseline
  The SF-36v2 is used to assess QoL. Consisting of 36 items, it assesses eight dimensions of health (dimensions of health (physical, performance limitations due to physical or emotional problems, intensity and discomfort due to pain, general health, vitality, social function and mental health). The global score range between 0 to 100. Higher scores indicate better the health-related QoL.
Change in QoL evaluated through SF-36v2 | 8 weeks after the beginning of the intervention
  The SF-36v2 is used to assess QoL. Consisting of 36 items, it assesses eight dimensions of health (dimensions of health (physical, performance limitations due to physical or emotional problems, intensity and discomfort due to pain, general health, vitality, social function and mental health). The global score range between 0 to 100. Higher scores indicate better the health-related QoL.
Change in QoL evaluated through SF-36v2 | 16 weeks after the beginning of the intervention
  The SF-36v2 is used to assess QoL. Consisting of 36 items, it assesses eight dimensions of health (dimensions of health (physical, performance limitations due to physical or emotional problems, intensity and discomfort due to pain, general health, vitality, social function and mental health). The global score range between 0 to 100. Higher scores indicate better the health-related QoL.
Change in QoL evaluated through SF-36v2 | 8 weeks after end of intervention
  The SF-36v2 is used to assess QoL. Consisting of 36 items, it assesses eight dimensions of health (dimensions of health (physical, performance limitations due to physical or emotional problems, intensity and discomfort due to pain, general health, vitality, social function and mental health). The global score range between 0 to 100. Higher scores indicate better the health-related QoL.

OTHER OUTCOMES:
Sociodemographic information gathered through the sociodemographic questionnaire | baseline
  Participants' answers in the sociodemographic questionnaire designed specifically for this study. It gathers information about gender, age, marital status, educational level, clinical diagnosis and will be administered to all participants.

CONTACTS AND LOCATIONS:
Overall Officials: Susana I Justo Henriques, Ph.D., Principal Investigator — Health Sciences Research Unit: Nursing (UICISA: E), Nursing School of Coimbra; Ana E Marques Castro, M.Sc., Principal Investigator — Cediara - Associação de Solidariedade Social de Ribeira de Fráguas; Enrique Pérez Sáez, Ph.D., Principal Investigator — National Reference Centre for Alzheimer's and Dementia Care, Imserso, Spain; Janessa O Carvalho, Ph.D., Principal Investigator — Bridgewater State University, Bridgewater, USA; Ana P Sargaço Mendes, MD, Principal Investigator — Centro Hospitalar do Baixo Vouga, Aveiro, Portugal
Locations (1):
- Cediara - Social Solidarity Association of Ribeira de Fráguas, Albergaria-a-Velha, Aveiro District, Portugal

IPD SHARING:
Plan to Share IPD: No